CLINICAL TRIAL: NCT06716697
Title: the Impact of Physical and Mental Fatigue on Balance
Status: Not yet recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Mohammed Torad, DR, Kafrelsheikh University
Other Study IDs: KFSIRB200-442
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Balance
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: physical and mental fatigue — physical and mental fatigue as a result of exposed to exams

SUMMARY:
Mental and physical Fatigue and overall fatigue will be collected based on Fatigue assessment scale while balance data will be obtained by recording mobile sensors in X, Y and Z directions when mobile placed on COG of the participants.

ELIGIBILITY:
Inclusion Criteria:

* patients from 18 to 24 years old

Exclusion Criteria:

* free of any mental disorders or major health issues in last year

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All young adults that work or have study load that affect their fatigue level
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 3 months
  Anteroposterior swaying

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Torad Torad, Principal Investigator — faculty of physical therapy
Locations (1):
- Faculy of Physical Therapy Kafrelshaikh University, Kafrelsheikh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes